CLINICAL TRIAL: NCT06130969
Title: Effects of Cervical Spine Retraction Exercise With and Without Diaphragmatic Breathing on Pain, Disability and Craniovertebral Angle in Forward Head Posture.
Brief Title: Effects of Cervical Spine Retraction Exercise With and Without Diaphragmatic Breathing in Forward Head Posture.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0155
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Forward Head Posture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Cervical Retraction exercise without diaphragmatic breathing along with baseline treatment
  Interventions: Other: Cervical Retraction Exercise; Other: Baseline Treatment
- Group B (Experimental): Cervical Retraction exercise with diaphragmatic breathing along with baseline treatment
  Interventions: Other: Cervical Retraction Exercise; Other: Diaphragmatic Breathing; Other: Baseline Treatment

INTERVENTIONS:
Other: Cervical Retraction Exercise — Participants will hold cervical retraction for 10 s up to 10 times. A break of 5 s will be provided per one movement and 30 s per one set. A total of three sets will be conducted. Therefore, the total exercise time will be <10 mints.
Other: Diaphragmatic Breathing — The diaphragmatic exercise will be performed in a supine position with 40° trunk flexion while holding 2.5 kg on the abdomen in the first 5 sessions and then 5 kg in the second 5 sessions. Participants will perform 3 sets with 10 repetitions at a ratio of one second of inspiration to two seconds of expiration, three sets of 15 repetitions at a ratio of two seconds of inspiration to four seconds of expiration, and three sets of 20 repetitions at a ratio of three seconds of inspiration to six seconds of expiration. The rest between rests will be 60 s.
  Arms: Group B
Other: Baseline Treatment — Hot fomentation will be given by applying cervical hot pack over the area in prone lying position for 10 mints and Isometric neck strengthening exercises (10 repetitions, each 5-second hold, 1 set) (20). • Nerve Stimulation (TENS) on the painful regions around the neck for 15 minutes with a TENS device. TENS parameters will be 150 μs square pulses with a frequency of 80 Hz.
  The intensity of the current will be adjusted to produce no contraction.
  • Posture education to keep upright posture during sitting.

SUMMARY:
This study aims to determine the effect of combining diaphragmatic exercises with cervical retraction exercise on pain, disability, active range of motions of cervical spine and craniovertebral angle in individuals with forward head posture.

DETAILED DESCRIPTION:
Forward head posture altering breathing pattern is one of the most common musculoskeletal deformity. Diaphragmatic exercises can reduce pain and disability levels, and correct forward head posture (FHP) in patients with neck discomfort.

In this randomized clinical trial, fifty two participants displaying forward head posture (FHP) will be randomly assigned to one of the two intervention groups: the Diaphragmatic Exercises and Cervical Retraction Exercise Combined Group or the Cervical Retraction Exercise Alone Group. Randomization will be performed using a convenient random sampling method via sealed opaque envelopes. Each participant will receive a total of twelve treatment sessions over a four-week period. The efficacy of the interventions will be assessed at the beginning (first session), conclusion (twelfth session), and two weeks after completing the sessions. Outcome measures, including pain intensity, disability levels, cervical range of motion, and craniovertebral angle (CVA), will be evaluated using the Numeric Pain Rating Scale (NPRS), Neck Disability Index (NDI), universal goniometer and Image J software, respectively. Data will be analyzed using Statistical Package for the Social Sciences (SPSS) software version 26. Normality of data will be assessed using the Kolmogorov-Smirnov test. For within-group comparisons, either repeated measures ANOVA or the Friedman test will be used. To compare changes between the groups, the independent t-test or Mann-Whitney U test will be applied, depending on the data distribution. The analysis of these outcome measures will provide valuable insights into the impact of the interventions on participants' symptoms and postural alignment.

ELIGIBILITY:
Inclusion Criteria:

* Primary complaint of neck pain (pain on the posterior part of the cervical spine to the beginning of the thoracic area with or without pain in the shoulder girdle)
* Age from 20 to 35 years
* Both gender
* CVA <49° (16)

Exclusion Criteria:

* Any serious pathology such as tumor
* Had history of whiplash injury within 3 months of the examination,
* Underwent prior surgery to the cervical spine
* Currently using muscle relaxation medication.
* Degenerative conditions
* Exhibited positive neurologic signs consistent with nerve root compression.
* Patients with a history of respiratory disease, such as repeated bronchitis, pneumonia, asthma, pulmonary lymph nodes, pleurisy, cured tuberculosis and others

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-02-10 (Estimated)

PRIMARY OUTCOMES:
Photogrammetry for Craniovertebral Angle (CVA) by image j software | 6 weeks
  CVA, can be measured using the lateral photos exposing C7 and the ear. The participants will maintain the natural head posture through the measurement method of self-balance posture. It is the angle made by the line that connects the seventh cervical spine with the tragus and the horizontal line of the seventh cervical spine in the sitting and standing positions. A CVA of <49° is characterized as FHP (3).
  Image J is an image processing and analysis program that can read both image file formats and raw formats. It can display, edit, analyze, process, store, and print images, as well as measure distances and angles.
Numeric pain rating scale (NPRS): | 6 weeks
  The NPRS is a subjective pain rating scale using an 11-point scale from 0 to 10, where 0 means 'no pain' and 10 means 'intolerable pain'. Participants select the whole number that best represents their level of pain.
Neck disability index (NDI): | 6 weeks
  that restricts the activities of daily living (ADL); it also helps to determine self- assessed disability. NDI has 10 domains covering pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Scores range from 0 to 50, with 50 being the greatest levels of dysfunction.
Goniometer for Cervical Range of motion (CROM) | 6 weeks
  Universal goniometer has fair inter-tester reliability ranging from 0.79-0.92. Validity of this tool is good i.e. 0.97-0.98 This tool is most commonly used in the clinical settings for evaluating joint ROM.

SECONDARY OUTCOMES:
Global rating of change (GRC) | 6 weeks
  GRC scale is used as an objective means to test the improvement of patient symptoms, to identify the intervention effect after treatment completion in clinical practice

CONTACTS AND LOCATIONS:
Overall Officials: Ali Raza, Principal Investigator — Riphah International University; Aneeqa Manzoor, Principal Investigator — Riphah International University
Locations (1):
- Chiropractor & Physio Pain Relief Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No